CLINICAL TRIAL: NCT03400787
Title: Latera Randomized Controlled Trial (RCT) - Latera® Absorbable Nasal Implant vs. Sham Control for Lateral Nasal Valve Collapse
Brief Title: Latera RCT - Latera vs. Sham Control for Lateral Nasal Valve Collapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spirox, Inc. (Industry)
Collaborators: New Arch Consulting (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP 04
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Nasal Valve Collapse; Nasal Breathing
Keywords: nasal airway obstruction; sham-control; Polylactide absorbable implant
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: Sham procedure participants will be allowed to crossover to receive Latera implants after the 3-month assessment if they continue to meet eligibility criteria. Crossover participants will be followed through 24 months post implant. Sham participants who do not crossover will be exited after the 3-month assessment.
Who Masked: Participant
Masking Description: Participants will be masked to treatment assignment through the 3-month assessment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Control Arm (Sham Comparator): Subjects in the Sham Control arm will undergo the same preoperative assessments as those in the Latera Treatment arm up to and including anesthesia for the implant, however, no implant will be placed.
  Crossover - Subjects will be unblinded after the 3-month assessment is complete. Eligible subjects in the Sham Control arm will be treated with the Latera Implant if they still meet all eligibility criteria. Follow up will continue to 24 months post-implant. Subjects who no longer meet the eligibility criteria will exit the study.
  Interventions: Device: Latera Implant
- Latera Treatment Arm (Experimental): Subjects in the active treatment arm will receive the Latera Implant using standard techniques. Follow up continues for 24 months post-implant.
  Interventions: Device: Sham Procedure

INTERVENTIONS:
Device: Latera Implant — Treatment with implant
  Arms: Sham Control Arm
Device: Sham Procedure — Sham procedure where the Latera delivery device is inserted but no implant delivered.
  Arms: Latera Treatment Arm

SUMMARY:
The primary objective of the LATERA RCT is to demonstrate the superiority of the Latera Implant to improve nasal breathing, compared with a Sham Control procedure.

DETAILED DESCRIPTION:
To evaluate the Latera Absorbable Nasal Implant (Latera Implant) Implant versus Sham Control in subjects with nasal valve collapse due to or primarily due to insufficient cartilaginous support of the lateral nasal wall.

ELIGIBILITY:
Subjects must meet the following criteria to be included in the study:

1. Adults aged 18 and above;
2. Understands and provides written informed consent;
3. Stated willingness to comply with all study procedures, post-treatment care and availability for the duration of the study follow up of 2 years;
4. In good general health as evidenced by medical history;
5. NOSE score ≥55;
6. Dynamic bi-lateral nasal wall insufficiency as confirmed by Positive Modified Cottle Maneuver;
7. Nasal and facial anatomy appropriate to receive the Latera Implant;
8. Documented failure of benefit after at least 4 weeks of conservative medical management, including, for example, antihistamines or nasal steroids, evidenced by lack of efficacy or tolerability.

Subjects meeting any one of the following criteria will be excluded for the study:

1. Unable to tolerate or not a candidate for procedures performed under local anesthesia;
2. Pathology other than lateral wall insufficiency (e.g. septal deviation, turbinate or adenoid hypertrophy, polyps, sinusitis, rhinitis) is the primary contributor to airway obstruction;
3. Requires or is anticipated to require any other concurrent nasal procedures (e.g. Functional Endoscopic Sinus Surgery (FESS), rhinoplasty, sinuplasty, septoplasty, or turbinate reduction) outside of the index procedure within 12 months after the index procedure;
4. FESS, sinuplasty, septoplasty, inferior turbinate reduction, or rhinoplasty within the past 6 months;
5. Any other rhinoplasty procedures are planned or planned usage of external dilators within 24 months after the index procedure;
6. Permanent nasal implant of any type (e.g. autologous, homologous, or synthetic graft) or dilator;
7. Presence of concomitant inflammatory or infectious conditions or unhealed wounds in the treatment area (e.g., vestibulitis, vasculitis, active acne),
8. Currently using chronic systemic steroids or recreational intra-nasal drugs;
9. Currently has cancerous or pre-cancerous nasal lesions, has had radiation in the treatment area, or is currently receiving chemotherapy;
10. History of a significant healing disorders including hypertrophic scarring, or keloid formation;
11. Poorly controlled diabetes mellitus;
12. Known or suspected allergy to PLA or other absorbable implant materials in the Latera Implant;
13. Severe obstructive sleep apnea (OSA) and cannot or is unwilling to refrain from continuous positive airway pressure (CPAP) for up to 2 weeks post-procedure based on expected healing needs and mask types, in agreement with the treating physician;
14. Female subjects, of child bearing potential, known or suspected to be pregnant or are lactating;
15. Any other presenting condition that, in the medical opinion of the investigator, would disqualify the subject from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Stolovitzky, MD, Principal Investigator — ENT of Georgia; Douglas Sidle, MD, Principal Investigator — Northwestern Facial Plastic Surgery
Locations (11):
- United States (11):
  - Sacramento ENT, Roseville, California
  - Breathe Clear Institute, Torrance, California
  - ENT of GA, Atlanta, Georgia
  - Chicago Nasal and Sinus Center, Chicago, Illinois
  - Michiana Sleep and ENT Solutions, South Bend, Indiana
  - Albany ENT & Allergy, Albany, New York
  - Piedmont ENT, Winston-Salem, North Carolina
  - Texas ENT Specialist, Houston, Texas
  - ENT Associates of Texas, McKinney, Texas
  - Texas Facial Plastics and ENT, San Antonio, Texas
  - Ogden Clinic, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stolovitzky P, Senior B, Ow RA, Mehendale N, Bikhazi N, Sidle DM. Assessment of bioabsorbable implant treatment for nasal valve collapse compared to a sham group: a randomized control trial. Int Forum Allergy Rhinol. 2019 Aug;9(8):850-856. doi: 10.1002/alr.22362. Epub 2019 Jun 21. PMID 31226238

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Control Arm: Subjects in the Sham Control arm will undergo the same preoperative assessments as those in the Latera Treatment arm up to and including anesthesia for the implant, however, no implant will be placed.
  Crossover - Subjects will be unblinded after the 3-month assessment is complete. Eligible subjects in the Sham Control arm will be treated with the Latera Implant if they still meet all eligibility criteria. Follow up will continue to 24 months post-implant. Subjects who no longer meet the eligibility criteria will exit the study.
  Latera Implant: Treatment
- Latera Treatment Arm: Subjects in the active treatment arm will receive the Latera Implant using standard techniques. Follow up continues for 24 months post-implant.
  Latera Implant: Treatment
Period: Overall Study
Arm/Group | Sham Control Arm | Latera Treatment Arm
Started | 66 | 71
3-Month Follow-up (1 participant randomized to sham inadvertently received an implant and was analyzed as treated.) | 64 | 63
Completed | 64 | 63
Not Completed | 2 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Unblinded before 3-month follow-upa- | 0 | 6

BASELINE CHARACTERISTICS:
Population: Participants with evaluable data for the primary endpoint at 3-month follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Control Arm | Latera Treatment Arm | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (13.5) | 50.9 (14.2) | 51.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 24 | 26 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 51 | 58 | 109
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 127
Baseline Nasal Obstruction Symptom Evaluation (NOSE) Score [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) is a validated patient-reported outcome assessment of 5 questions relating to nasal obstruction (congestion, obstruction, trouble breathing through the nose, trouble sleeping, unable to breath through the nose during exercise/exertion. Each question is rated on a Likert scale of 0 (no problem) to 4 (severe problem). The sum of the scores is multiplied by 5 to result in a total score that ranges from 0 to 100.
  units on a scale | 77.7 (15.1) | 77.4 (13.1) | 77.6 (14.1)

OUTCOME MEASURES:

1. Primary Outcome: NOSE Responder Rate
Description: The primary endpoint of the study is the NOSE Responder Rate, assessed 3 months post-procedure in the per-protocol population of the Latera and Sham arms. The Nasal Obstruction Symptom Evaluation (NOSE) is a validated patient-reported outcome assessment of 5 questions relating to nasal obstruction (congestion, obstruction, trouble breathing through the nose, trouble sleeping, unable to breath through the nose during exercise/exertion. Each question is rated on a Likert scale of 0 (no problem) to 4 (severe problem). The sum of the scores is multiplied by 5 to result in a total score that ranges from 0 to 100. NOSE scores can also be categorized as mild (5-25), moderate (30-50), severe (55-75), and extreme (80-100). A NOSE responder is defined as a participant with at least 1 NOSE class improvement or at least 20% total NOSE score reduction.
Time Frame: 3 months postprocedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control Arm | Latera Treatment Arm
Number analyzed (Participants) | 64 | 63
Participants | 35 | 52
Statistical Analysis 1: Comparison: Sham Control Arm vs Latera Treatment Arm; Null hypothesis is that the responder rate for the Latera implant treatment was not superior to the sham treatment. A maximum sample size of 124 evaluable subjects is required for 90% power and preserving a 2.5% (one-sided) type I error rate; Test type: Superiority; p = 0.0001, t-test, 1 sided — p<0.025 indicates statistical significance

2. Secondary Outcome: Responder Rate
Description: Responder Rate at 7 days, 30 days, and 6, 12, 18 and 24 months will be assessed
Time Frame: 7 days, 30 days, and 6, 12, 18 and 24 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events reported from procedure through 3-month follow-up.
Arm/Group | Sham Control Arm | Latera Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/64 | 3/63
Other Adverse Events (participants affected / at risk) | 0/64 | 5/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control Arm (N=64) | Latera Treatment Arm (N=63)
Liver cancer (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related to study device or procedure
Degenerative disc disease/stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not related to study device or procedure
Death (General disorders) | 1 (1) | 0 (0) — Unknown cause of death. Not related to study device or procedure
Severe hypertension (General disorders) | 0 (0) | 1 (1) — Not related to study device or procedure
Orthopedic surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Right knee surgery. Not related to study device or procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Control Arm (N=64) | Latera Treatment Arm (N=63)
Implant extrusion/migration (Product Issues) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT03400787/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03400787/SAP_001.pdf